CLINICAL TRIAL: NCT00552097
Title: Effect of Combination Ezetimibe and High-Dose Simvastatin vs Simvastatin Alone on the Atherosclerotic Process in Subjects With Heterozygous Familial Hypercholesterolemia (The ENHANCE Trial)
Brief Title: Effect of Ezetimibe Plus Simvastatin Versus Simvastatin Alone on Atherosclerosis in the Carotid Artery (ENHANCE)(P02578)
Acronym: ENHANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P02578
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Atherosclerosis; Hypercholesterolemia; Hyperlipoproteinemia Type II
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — Ezetimibe; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EZ/Simva (Experimental)
  Interventions: Drug: ezetimibe (plus simvastatin)
- Placebo/Simva (Placebo Comparator)
  Interventions: Drug: placebo (plus simvastatin)

INTERVENTIONS:
Drug: ezetimibe (plus simvastatin) — oral tablets; ezetimibe 10 mg (plus simvastatin 80 mg) once daily for 24 months
  Other Names: ZETIA; VYTORIN; SCH 58235; SCH 465981
  Arms: EZ/Simva
Drug: placebo (plus simvastatin) — tablets; placebo to match ezetimibe 10 mg (plus simvastatin 80 mg) once daily for 24 months
  Arms: Placebo/Simva

SUMMARY:
The purpose of the study is to determine whether ezetimibe plus simvastatin will be more effective than simvastatin alone in preventing progression of atherosclerosis of the inner layer of the carotid artery.

ELIGIBILITY:
Inclusion Criteria:

* Genotype-confirmed heterozygous familial hypercholesterolemia with written documentation of the genetic diagnosis at the time of screening and LDL-C >=210 mg/dL (5.43 mmol/L), or clinical diagnosis of heterozygous familial hypercholesterolemia, defined as LDL-C >=210 mg/dL (5.43 mmol/L) and at least one of the following:

  * tendinous xanthoma
  * child <18 years of age with hypercholesterolemia (LDL-C >159 mg/dL (4.11 mmol/L)
  * has a sibling with hypercholesterolemia (LDL-C >190 mg/dL [4.91 mmol/L]) and tendinous xanthoma
  * family history with an LDL-C value distribution pattern compatible with dominant autosomal transmission and at least one relative presenting fasting total cholesterol values >348 mg/dL (9.0 mmol/L) after exclusion of secondary causes of dyslipidemia
* LDL-C >=210 mg/dL (5.43 mmol/L) 1 week before randomization
* plasma triglyceride level <=400 mg/dL (4.52 mmol/L)

Exclusion Criteria:

* pregnancy or any other situation, condition, or illness that, in the opinion of the investigator, may interfere with optimal participation in the study
* presence of an apolipoprotein B gene mutation with confirmed absence of an LDL receptor mutation in either allele
* undergoing LDL-apheresis or plasma apheresis
* unsuitable plaque or artery morphology
* use of certain drugs, foods, or other agents known to alter cholesterol levels or to cause pharmacokinetic interactions with either ezetimibe or simvastatin

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2002-06-01 (Actual); Primary Completion 2006-04-25 (Actual); Study Completion 2006-04-25 (Actual)

PRIMARY OUTCOMES:
Change in ultrasound-determined average carotid artery intima-media thickness (IMT) on a per subject basis between baseline and endpoint. | 24 months

SECONDARY OUTCOMES:
Proportion of subjects with a reduction in ultrasound-determined average carotid artery IMT between baseline and endpoint. | 24 months
Change in ultrasound-determined maximum carotid artery IMT on a per subject basis between baseline and endpoint. | 24 months
Proportion of subjects developing new carotid artery plaques between baseline and endpoint. | 24 months
Change in ultrasound-determined average carotid artery plus average common femoral artery IMT on a per subject basis between baseline and endpoint. | 24 months

REFERENCES:
- [Background] Kastelein JJ, Sager PT, de Groot E, Veltri E. Comparison of ezetimibe plus simvastatin versus simvastatin monotherapy on atherosclerosis progression in familial hypercholesterolemia. Design and rationale of the Ezetimibe and Simvastatin in Hypercholesterolemia Enhances Atherosclerosis Regression (ENHANCE) trial. Am Heart J. 2005 Feb;149(2):234-9. doi: 10.1016/j.ahj.2004.06.024. PMID 15846260
- [Derived] Kastelein JJ, Akdim F, Stroes ES, Zwinderman AH, Bots ML, Stalenhoef AF, Visseren FL, Sijbrands EJ, Trip MD, Stein EA, Gaudet D, Duivenvoorden R, Veltri EP, Marais AD, de Groot E; ENHANCE Investigators. Simvastatin with or without ezetimibe in familial hypercholesterolemia. N Engl J Med. 2008 Apr 3;358(14):1431-43. doi: 10.1056/NEJMoa0800742. Epub 2008 Mar 30. PMID 18376000